CLINICAL TRIAL: NCT06566313
Title: An Open-label Study on the Clinical Efficacy of tDCS Intervention in PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHMU-tDCS-PD
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Transcranial Direct Current Stimulation; Parkinson Disease; Primary Left Motor Cortex
Keywords: Transcranial Direct Current Stimulation; Parkinson Disease; primary left motor cortex
MeSH Terms: conditions — Parkinson Disease | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tDCS group (Experimental): a course of tDCS treatment is performed for 10 days
  Interventions: Behavioral: transcranial Direct Current Stimulation

INTERVENTIONS:
Behavioral: transcranial Direct Current Stimulation — On the basis of conventional anti-PD drugs, the left M1 region (based on the C3 coordinates of EEG 10-20 system and the surrounding FC1, FC5, CP1, CP5 coordinates) was treated with cathodic tDCS. The electrical stimulation intensity was 2.0mA, the treatment time was 20min, and the treatment lasted for 10 days.

SUMMARY:
To demonstrate that intervention targeting the primary motor area (M1) using transcranial Direct Current Stimulation can improve sleep symptoms in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Rapid eye movement sleep behavior disorder (RBD) is one of the most common accompanying symptoms of Parkinson's disease (PD). PD-RBD patients have more severe clinical manifestations, require larger drug doses, and have more non-motor symptoms. Although several strategies using transcranial direct current stimulation (tDCS) have been investigated for the treatment of sleep disorders, the efficacy of high-definition tDCS (HD-tDCS) in PD-RBD patients remains unclear.

We conducted an open-label study using the RBD-SQ to identify individuals with possible RBD (pRBD), and recruiting the patients at the First Affiliated Hospital of Anhui Medical University to receive cathodal HD-tDCS intervention. On the basis of conventional anti-PD drugs, cathodal HD-tDCS treatment was performed on the left M1 area once a day for 20 minutes, and the treatment was continued for 10 days. The International Movement Disorders Society Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), the Hoehn & Yahr staging scale (H&Y), REM Sleep Behavior Disorder Screening Questionnaire (RBDSQ), RBD Screening Questionnaire Hong Kong (RBDSQ- HK), Pittsburgh sleep quality index (PSQI), Epworth Sleepiness Scale (ESS), and Parkinson disease sleep scale (PDSS) were assessed on intervention Day 1 and Day 10, and clinical efficacy was evaluated by comparing the scale scores before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of PD was determined by neurologists with rich clinical work experience, and was in line with the diagnostic criteria for Parkinson's disease in China (2016 edition).
2. The total score of RBD Screening Questionnaire (RBDSQ) is ≥6 points.
3. All patients took the drug stably and had no history of drug adjustment within 2 months before treatment. The test was conducted 2 hours after taking the drug.
4. Good compatibility, with a certain degree of compliance;
5. Normal mental condition, able to cooperate with behavioral tests and transcranial electrical stimulation treatment;

Exclusion Criteria:

1. The patient has a metal object or skull brace device or any similar metal object on the scalp;
2. Head tremor or limb shaking is so severe that it is difficult to calmly receive treatment;
3. The presence of other serious mental illness (such as major depression, psychosis or obsessive-compulsive disorder, physical illness or a history of substance abuse);
4. Have a head injury, stroke or other neurological disorder;
5. The diagnosis of PD dementia is difficult to complete the assessment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
RBD Screening Questionnaire | baseline; day 10
  The RBD Screening Questionnaire (RBDSQ) is the most widely used tool over the past decade and includes 13 yes-or-no questions regarding the presence of move- ments and dream-enacting behaviours during sleep(maximum total score 13 points) .

SECONDARY OUTCOMES:
REM sleep behavior disorder questionnaire-Hong Kong | baseline; day 10
  The RBDQ-HK questionnaire is a self-administered (by patient and/or bed partner) questionnaire comprising 13 questions per- taining to various clinical features of RBD as defined by the Inter- national Classification of Sleep Disorders (ICSD-II).The total RBD score was calcu- lated by the sum of the scores of all lifetime items and recent 1- year frequency items. The total RBD score has a range from 0 to 100.
Pittsburgh sleep quality index | baseline; day 10
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a l-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.
EPworth Sleepiness Scale | baseline; day 10
  The Epworth sleepiness scale (ESS) is asimple, self-administered questionnaire which is shown to provide a measurement of the subject's genera1level of daytime sleepiness.
Parkinson disease sleep scale | baseline; day 10
  The PDSS is a visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance.This is the description of a simple bedside screening instrument for evaluation of sleep disturbances in Parkinson's disease.
Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale | baseline; day 10
  The MDS-UPDRS is used to diagnose Parkinson's disease and assess the severity of symptoms, which is based on three major motor manifestations. Parkinson's disease is defined as bradykinesia with resting tremor, rigidity, or both.

CONTACTS AND LOCATIONS:
Overall Officials: Panpan Hu, MD, Principal Investigator — The First Affiliated Hospital of Anhui Medical University
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No